CLINICAL TRIAL: NCT02829385
Title: A Phase II Clinical Trial Study on Apatinib and XELOX Combination Regimen in the First-line Treatment of End-stage Colorectal Cancer Patients
Brief Title: Clinical Study of Apatinib and XELOX Combination Regimen to Treat Colorectal Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shoucheng Ma (Other)
Responsible Party: Sponsor-Investigator, Shoucheng Ma, director of cancer center, LanZhou University
Organization: LanZhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LZU-123
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Neoplasms
Keywords: Apatinib; XELOX Regimen; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apatinib combined treatment group (Experimental): Apatinib Mesylate Tablets 500 mg P.O.d1-21 and XELOX (oxaliplatin 130mg/㎡ i.v. d1, capecitabine 1000mg P.O. d1-d14)
  Every 3-week time is a cycle until PD or intolerance of drug toxicity occurs.
  Interventions: Drug: Apatinib and XELOX combined treatment group

INTERVENTIONS:
Drug: Apatinib and XELOX combined treatment group — Apatinib Mesylate Tablets 500 mg P.O.d1-21 and XELOX (oxaliplatin 130mg/㎡ i.v. d1, capecitabine 1000mg P.O. d1-d14)
  Every 3-week time is a cycle until PD or intolerance of drug toxicity occurs.
  Other Names: Apatinib combined treatment group

SUMMARY:
This study makes an observation over the objective response rate of Apatinib and XELOX combination regimen in the first-line treatment of metastatic colorectal cancer. All the participants will receive the treatment of Apatinib and XELOX combination regimen.

DETAILED DESCRIPTION:
XELOX chemotherapy is an effective therapy for metastatic colorectal cancer as first-line treatment.

Apatinib is a small-molecule tyrosine kinase inhibitor (TKI) that highly selectively binds to and strongly inhibits vascular endothelial growth factor receptor 2 (VEGFR-2), with a decrease in VEGF-mediated endothelial cell migration, proliferation, and tumor microvascular density. A phase II trail of Apatinib has been demonstrated that Apatinib is safe to treat the metastatic colorectal cancer and the disease control rate can reach 50%.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable colorectal cancer confirmed by histological means with measurable indication（a minimum size of 10mm by spiral CT scan，which meets the criteria of RECIST 1.1）.
* Time interval traced back to the latest administration of xelox and folfox combination must be no less than 1 year.
* age range: ≥18 and ≤75.
* ECOG PS scale 0 or 1；expected survival time ≥12 weeks.
* Sufficient blood function：absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥80×109/L and hemoglobin≥9g/dL.
* Sufficient hepatic function：total bilirubin ≤1.5 times upper normal limit(ULN), AST ≤2.5 times ULN, ALT ≤2.5 times ULN and AKP ≤5 times ULN.

  *AST,ALT relevant criteria alters into AST ≤5 times ULN and ALT ≤5 times ULN if with hepatic metastasis.
* sufficient renal function: serum creatinin ≤ULN, creatinine clearance rate ≥60 mL/min
* Female patients under age 50 with complete uterus must be tested negative for pregnancy within 28 days before enrollment (except for those who suffered amenorrhea for more than 24 months). If the pregnancy test was carried out more than 7 days before the first administration, then the urine pregnancy test is required for validation. (within the 7-day interval before administration)
* Informed consent subscription. (The consent should be approved by independent Ethics Committee, and signed by patients before any substantial trial is initiated.)

Exclusion Criteria:

* Have got other malignant tumors within last 5 years, excluding basal cell skin cancer and cervical carcinoma in situ that has already been cured.
* With evidence of CNS metastasis, even if the treatment had been carried out before, patients with doubts of CNS metastasis should be conducted MRI or enhanced CT scan on within 28 days before enrollment for ruling out.
* AST ≤2.5 times ULN and/or ALT ≤2.5 times ULN
* Had been treated with chemotherapy for last 12 months
* Had been treated with radiotherapy (except for palliative radiotherapy with evaluable focus outside radiotherapy field on purpose of alleviating pains)
* With any uncontrolled systemic disease, including active infection, hypertension without treatment, diabetes mellitus, angina pectoris, congestive heart failure, myocardial infarction, severe arrhythmia requires treatment and hepatic/renal/metabolic diseases
* Taking experimental treatment from another clinical trial study.
* Being allergic to any relevant chemotherapy drug.
* With evidence-proved other diseases, neural or metabolic disorders, physical or lab examination abnormalities, which might be contraindication of study drugs or leading to treating-related lethal complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 9 months
  ORR=complete response (CR) + partial response (PR) .And expected ORR is 0.55.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | up to 2 years
  time from randomization to documented progressive disease or death due to any cause, whichever occurs first
Overall Survival (OS) | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Da Zhao, Bachelor, Study Chair — Cancer Center of the First Hospital of Lanzhou University
Locations (1):
- Cancer Cnter,The First Hospital of Lanzhou University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- [Result] Tabernero J, Van Cutsem E, Lakomy R, Prausova J, Ruff P, van Hazel GA, Moiseyenko VM, Ferry DR, McKendrick JJ, Soussan-Lazard K, Chevalier S, Allegra CJ. Aflibercept versus placebo in combination with fluorouracil, leucovorin and irinotecan in the treatment of previously treated metastatic colorectal cancer: prespecified subgroup analyses from the VELOUR trial. Eur J Cancer. 2014 Jan;50(2):320-31. doi: 10.1016/j.ejca.2013.09.013. Epub 2013 Oct 16. PMID 24140268
- [Result] Kara O, Duman BB, Kara B, Erdogan S, Parsak CK, Sakman G. Analysis of PTEN, VEGF, HER2 and P53 status in determining colorectal cancer benefit from bevacizumab therapy. Asian Pac J Cancer Prev. 2012;13(12):6397-401. doi: 10.7314/apjcp.2012.13.12.6397. PMID 23464465
- [Result] Custodio A, Barriuso J, de Castro J, Martinez-Marin V, Moreno V, Rodriguez-Salas N, Feliu J. Molecular markers to predict outcome to antiangiogenic therapies in colorectal cancer: current evidence and future perspectives. Cancer Treat Rev. 2013 Dec;39(8):908-24. doi: 10.1016/j.ctrv.2013.02.004. Epub 2013 Mar 16. PMID 23510598
- [Result] Bruera G, Cannita K, Giordano AV, Vicentini R, Ficorella C, Ricevuto E. Effectiveness and safety of intensive triplet chemotherapy plus bevacizumab, FIr-B/FOx, in young-elderly metastatic colorectal cancer patients. Biomed Res Int. 2013;2013:143273. doi: 10.1155/2013/143273. Epub 2013 Nov 6. PMID 24307987
- [Result] Sclafani F, Cunningham D. Bevacizumab in elderly patients with metastatic colorectal cancer. J Geriatr Oncol. 2014 Jan;5(1):78-88. doi: 10.1016/j.jgo.2013.08.006. Epub 2013 Sep 20. PMID 24484722
- [Result] Naeim A, Ward PR, Wang HJ, Dichmann R, Liem AK, Chan D, Patel R, Hu EH, Tchekmedyian NS, Wainberg ZA, Hecht JR. A phase II trial of frontline capecitabine and bevacizumab in poor performance status and/or elderly patients with metastatic colorectal cancer. J Geriatr Oncol. 2013 Oct;4(4):302-9. doi: 10.1016/j.jgo.2013.05.001. Epub 2013 Jun 7. PMID 24472472
- [Result] Simkens LH, van Tinteren H, May A, ten Tije AJ, Creemers GJ, Loosveld OJ, de Jongh FE, Erdkamp FL, Erjavec Z, van der Torren AM, Tol J, Braun HJ, Nieboer P, van der Hoeven JJ, Haasjes JG, Jansen RL, Wals J, Cats A, Derleyn VA, Honkoop AH, Mol L, Punt CJ, Koopman M. Maintenance treatment with capecitabine and bevacizumab in metastatic colorectal cancer (CAIRO3): a phase 3 randomised controlled trial of the Dutch Colorectal Cancer Group. Lancet. 2015 May 9;385(9980):1843-52. doi: 10.1016/S0140-6736(14)62004-3. Epub 2015 Apr 7. PMID 25862517
- [Result] Kiss I, Bortlicek Z, Melichar B, Poprach A, Halamkova J, Vyzula R, Dusek L, Buchler T. Efficacy and toxicity of bevacizumab on combination with chemotherapy in different lines of treatment for metastatic colorectal carcinoma. Anticancer Res. 2014 Feb;34(2):949-54. PMID 24511038
- [Result] Kishiki T, Ohnishi H, Masaki T, Ohtsuka K, Ohkura Y, Furuse J, Watanabe T, Sugiyama M. Overexpression of MET is a new predictive marker for anti-EGFR therapy in metastatic colorectal cancer with wild-type KRAS. Cancer Chemother Pharmacol. 2014 Apr;73(4):749-57. doi: 10.1007/s00280-014-2401-4. Epub 2014 Feb 6. PMID 24500024
- [Result] Peeters M, Oliner KS, Price TJ, Cervantes A, Sobrero AF, Ducreux M, Hotko Y, Andre T, Chan E, Lordick F, Punt CJ, Strickland AH, Wilson G, Ciuleanu TE, Roman L, Van Cutsem E, He P, Yu H, Koukakis R, Terwey JH, Jung AS, Sidhu R, Patterson SD. Analysis of KRAS/NRAS Mutations in a Phase III Study of Panitumumab with FOLFIRI Compared with FOLFIRI Alone as Second-line Treatment for Metastatic Colorectal Cancer. Clin Cancer Res. 2015 Dec 15;21(24):5469-79. doi: 10.1158/1078-0432.CCR-15-0526. Epub 2015 Sep 4. PMID 26341920
- [Result] Douillard JY, Oliner KS, Siena S, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Williams R, Rong A, Wiezorek J, Sidhu R, Patterson SD. Panitumumab-FOLFOX4 treatment and RAS mutations in colorectal cancer. N Engl J Med. 2013 Sep 12;369(11):1023-34. doi: 10.1056/NEJMoa1305275. PMID 24024839